CLINICAL TRIAL: NCT00130975
Title: Candesartan in the Prevention of Relapsing Atrial Fibrillation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asker & Baerum Hospital (Other)
Collaborators: Helse Ost (Unknown); Ullevaal University Hospital (Other); AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPRAF
Record Dates: First submitted 2005-08-16; First posted 2005-08-17 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2007-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation.; Cardioversion.; Recurrence.; Candesartan.
MeSH Terms: conditions — Atrial Fibrillation; Recurrence | interventions — candesartan

INTERVENTIONS:
Drug: Candesartan

SUMMARY:
The purpose of this study is to test the hypothesis that treatment with the angiotensin II type 1 receptor antagonist candesartan may reduce the recurrence rate of atrial fibrillation after electrical cardioversion.

DETAILED DESCRIPTION:
Background: The most effective procedure to restore sinus rhythm in patients with persistent atrial fibrillation (AF) is electrical cardioversion, but AF recurs in 60-80% of the patients during the first year. AF is associated with electrical and anatomical remodelling of the atria, and angiotensin II is involved in the remodelling process. Studies have indicated that the angiotensin II type 1 receptor antagonist candesartan may counteract both electrical and anatomical remodelling induced by AF. The investigators therefore hypothesised that treatment with candesartan may reduce the recurrence rate of AF after electrical cardioversion.

Study design: 171 patients with persistent AF scheduled for electrical cardioversion are randomised in a double blind, placebo-controlled study. The patients receive tablets of candesartan 8 mg or matching placebo once daily for 3-6 weeks before cardioversion, and candesartan 16 mg or matching placebo once daily for 6 months after cardioversion. The study medication is discontinued if electrical cardioversion is unsuccessful or if AF recurrence is documented. Primary endpoint is recurrence of AF. Clinical, electrocardiographic, echocardiographic and biochemical markers will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrial fibrillation, diagnosed electrocardiographically, of more than 48 hours duration in whom direct current (DC) cardioversion is planned.

Exclusion Criteria:

* Patients with a history of known hypersensitivity or contraindication to any angiotensin II receptor blocker or any angiotensin-converting enzyme (ACE) inhibitor.
* Patients currently receiving an ACE inhibitor or angiotensin II antagonist because of heart failure or other strong indication.
* Patients currently receiving any antiarrhythmic medication including sotalol. Other beta-blockers will not be regarded as specific antiarrhythmic agents.
* Significant renal artery stenosis and any medical condition in which administration of a vasodilator is contraindicated; serum creatinine > 225 micromol/L; or serum potassium > 5.5 mmol/L; or serum sodium < 128 mmol/L.
* Patients with severe hepatic dysfunction.
* Life-limiting disease or substance abuse which may affect participation.
* Patients unwilling to participate.
* Patients who have previously undergone DC cardioversion for atrial fibrillation within the last month.
* Thyrotoxicosis.
* Patients with a systolic blood pressure of < 100 mm Hg.
* Hypertensive patients requiring intensified treatment prior to DC cardioversion.
* Pregnancy or lactation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2001-04; Study Completion 2005-09

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation

SECONDARY OUTCOMES:
Time to recurrence of atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Arnljot Tveit, MD, Principal Investigator — Asker & Baerum Hospital
Locations (2):
- Norway (2):
  - Ulleval University Hospital, Oslo
  - Asker & Baerum Hospital, Rud

REFERENCES:
- [Result] Tveit A, Grundvold I, Olufsen M, Seljeflot I, Abdelnoor M, Arnesen H, Smith P. Candesartan in the prevention of relapsing atrial fibrillation. Int J Cardiol. 2007 Aug 9;120(1):85-91. doi: 10.1016/j.ijcard.2006.08.086. Epub 2006 Nov 17. PMID 17113170
- [Derived] Horjen AW, Seljeflot I, Berge T, Smith P, Arnesen H, Tveit A. Effect of sinus rhythm restoration on markers of thrombin generation in atrial fibrillation. Thromb J. 2017 Dec 28;15:30. doi: 10.1186/s12959-017-0153-1. eCollection 2017. PMID 29299030